CLINICAL TRIAL: NCT01793844
Title: A Prospective , Multicenter, Randomized Phase III Study of Improving the Efficacy of Treatment in Diffused Large B Cell Lymphoma Patients
Brief Title: A Study of Improving the Efficacy of Treatment in Diffused Large B Cell Lymphoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Tongyu Lin, vice chairman of department of medical oncology, Sun Yat-sen University
Other Study IDs: CSWOG0001
Record Dates: First submitted 2008-12-24; First posted 2013-02-18 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: diffuse large B cell lymphoma; DFS; OS
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- A (R-CHOP21): CHOP combined with Rituximab regimen（R-CHOP21）
  Treatment Arm A(R-CHOP21): Rituximab 375mg/m2 for injection on day1; cyclophosphamide(C), 750mg/m2 for injection on day2; doxorubicin(H), 50mg/m2 for injection on day2; and Vincristine(O), 1.4mg/m2 for injection on day2, prednisone(P) 60mg/m2 orally on days 2 to 6. The therapy was repeated every 21 days for a total of 6 cycles.
- B (CHOP14): Biweekly CHOP regimen （CHOP14） Treatment Arm B (CHOP14): cyclophosphamide(C), 750mg/m2 for injection on day1; doxorubicin(H), 50mg/m2 for injection on day1; and Vincristine(O), 1.4 mg/m2 for injection on day1, prednisone(P) 60mg/m2 orally on days 1 to 5. The therapy was repeated every 14 days for a total of 6 cycles.PS: G-CSF 1.0-2ug/kg/ d for subcutaneous injections will be administered on day 6 for a total use of 6-8 days.
- C （R-CHOP14): Biweekly CHOP combined with Rituximab regimen（R-CHOP14） Treatment Arm C (R-CHOP14): Rituximab 375mg/m2 for injection on day1; cyclophosphamide(C), 750mg/m2 for injection on day2; doxorubicin(H), 50mg/m2 for injection on day2; and Vincristine(O), 1.4mg/m2 for injection on day2, prednisone(P),60mg/m2 orally on days 2 to 6. The therapy was repeated every 14 days for a total of 6 cycles.PS: G-CSF 1.0-2ug/kg/ d for subcutaneous injections will be administered on day 7 for a total use of 6-8 days patients with bulky disease or extranodal lesion wil be received radiotherapy after finishing the chemotherapy.

SUMMARY:
This is a prospective , open, multicenter, randomized phase Ⅲ study. The investigators planed to include 732 untreated CD20 positive diffused large B cell lymphoma adults,to random to R-CHOP21, CHOP14 , R-CHOP14 regimen groups after signature the informed consents. The patients will receive safety assessment every cycles, and efficacy evaluation every 2 cycles. Every-two-months follow up will be received after finishing the treatment.

DETAILED DESCRIPTION:
This is a prospective , open, multicenter, randomized phase Ⅲ study. We planed to include 732 untreated CD20 positive diffused large B cell lymphoma adults,to random to R-CHOP21, CHOP14 , R-CHOP14 regimen groups after signature the informed consents. The patients will receive safety assessment every cycles, and efficacy evaluation every 2 cycles. Every-two-months follow up will be received after finishing the treatment.

* randomization Subjects will be randomly assigned to 1 of 3 treatment groups based on a computer-generated randomization schedule prepared before the study.
* Dosage and administration

  * Treatment Arm A(R-CHOP21): Rituximab 375mg/m2 for injection on day1; cyclophosphamide(C), 750mg/m2 for injection on day2; doxorubicin(H), 50mg/m2 for injection on day2; and Vincristine(O), 1.4mg/m2 for injection on day2, prednisone(P) 60mg/m2 orally on days 2 to 6. The therapy was repeated every 21 days for a total of 6 cycles.
  * Treatment Arm B (CHOP14): cyclophosphamide(C), 750mg/m2 for injection on day1; doxorubicin(H), 50mg/m2 for injection on day1; and Vincristine(O), 1.4 mg/m2 for injection on day1, prednisone(P) 60mg/m2 orally on days 1 to 5. The therapy was repeated every 14 days for a total of 6 cycles.PS: G-CSF 1.0-2ug/kg/ d for subcutaneous injections will be administered on day 6 for a total use of 6-8 days.
  * Treatment Arm C (R-CHOP14): Rituximab 375mg/m2 for injection on day1; cyclophosphamide(C), 750mg/m2 for injection on day2; doxorubicin(H), 50mg/m2 for injection on day2; and Vincristine(O), 1.4mg/m2 for injection on day2, prednisone(P),60mg/m2 orally on days 2 to 6. The therapy was repeated every 14 days for a total of 6 cycles.PS: G-CSF 1.0-2ug/kg/ d for subcutaneous injections will be administered on day 7 for a total use of 6-8 days patients with bulky disease or extranodal lesion wil be received radiotherapy after finishing the chemotherapy.
* Study evaluations

  * Criteria for response categories Tumour response will be evaluated according to the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas(1998)
  * Efficacy Criteria Disease-free survival Disease-free survival for patients in CR or CRu is measured from the first assessment that documents that response to the date of disease progression or the most recent follow-up visit time. Response rate Response rate is defined as the proportion of subjects who achieve CR/Cru and PR relative to the total population.Overall survival Overall survival is measured from entry onto the study until death from any cause, or the most recent follow-up visit date
  * Scheduling of tumour assessments Baseline total tumour burden must be assessed within a maximum of 21 days before first dose of treatment.Follow-up tumour evaluations will be performed during the last week of every 2nd cycle. After finishing the therapies, tumor evaluation will be performed every 3 months in the first and second years,following every 6 months after 2 years. tumour assessments may be performed by CT/MRI for the internal organs lesion. In case of clinically measurable superficial lesions, accurate evidence should be performed in the original records.
* Clinical Safety Assessments

The following, safety, assessments and procedures will be performed according to the schedule of assessments:

* A complete medical history (including demographics, smoking history, cancer/treatment history) will be performed at screening.
* Physical examination
* ECG
* Weight
* Blood pressure
* heart rate
* respiratory rate
* ECOG Score
* Infection signs Adverse Events and Serious Adverse Events (SAEs) reported according to NCI-CTC criteria. Patients will be assessed for adverse events at each clinical visit and as necessary throughout the study.

  * Laboratory Safety Assessments

The following will be completed according to the schedule of assessments:

* Hæmoglobin
* Haematocrit
* Leucocytes
* Neutrophils
* Platelets
* Serum electrolytes ( K+, Ca++)
* Serum chemistries (Total bilirubin, ALT [SGPT], AST [SGOT], total protein, albumin, LDH, alkaline phosphatase, urea [BUN], serum creatinine, creatinine clearance).
* Dipstick urinalysis. In case of a significant finding, a microscopic urinalysis should be performed.

Note:Adverse Events and Serious Adverse Events (SAEs) reported according to NCI-CTC criteria(Version 3.0)Patients will be assessed for adverse events at each clinical visit and as necessary throughout the study.

* Follow-up Patients on the study should be reassessed after completion of treatment at a minimum of every 3 months for 2 years, then every 6 months until the completion of the study.assessment content at follow-up visits should include history, physical examination ,blood picture, Urinalysis,liver and kidney function and tumor assessments.
* Statistical analyzes The proposed regimen was to be considered worthy for additional investigation in this patient population if a disease control rate of 15% or greater. The total sample size will be about 636 patients (to collect 732 evaluable patients, considering a drop-out rate of around 10%, each group number: 244). Treatment duration was defined as days from the first day of drug administration to the last regulated rest day of the final cycle.,Primary objective is disease free survival. Secondary objectives are response rate, safety and 5-year overall survival.

Response rate is estimated using the binomial probability and exact 95% confidence intervals (CIs) were provided. disease free survival and overall survival curves are estimated using Kaplan-Meier methodology.

Adverse events and laboratory tests graded according to the NCI-CTC AE(Version 3.0).Adverse events will be assigned preferred terms and categorized into body systems according to the MEDDRA classification of the WHO terminology.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤70 years old.
* Histological documented untreated CD20(+) diffused large B cell lymphoma.
* Measurable disease and evaluable lesion.
* Never previously treated with radiotherapy, chemotherapy or surgery for malignant disease.
* Normal Haematological,liver and kidney function (Neutrophil count ≥ 1.5 × 109/L ,hemoglobin ≥ 100g/L,platelets ≥ 100 × 109/L)
* ECOG Performance status 0-3,Life expectancy of at least 3 months.
* Without history of another malignancy
* Without any conflict serious systemic disease
* Without any accompany treatment(including steroids drugs)
* Subjects must have signed and informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Female subjects must be practicing and effective methods of birth control for at least 6 months throughout and after study; and have a negative serum β-hCG pregnancy test at screening.

Exclusion Criteria

* Patients with prior clinical study within 3 months.
* Secondary lymphoma induced by chemotherapy or radiotherapy for another malignancy
* Transformed lymphoma
* Primary central nervous system lymphoma or primary testis lymphoma
* History of allergic reaction to any ectogenic proteins
* Prior treatment for lymphoma .
* History of another malignancy
* Neutrophil count < 1.0× 109/L ,hemoglobin < 90g/L,platelets < 90 × 109/L,concurrent treatment with systemic antibiotic or antiviral drug for active infection.
* Decompensated heart failure, dilated cardiomyopathy, coronary artery disease with depression of ST-T for electrocardiogram, myocardial infarction within 6 months
* Serious infective or organic disease
* Kidney dysfunction not related to lymphoma(Creatinine clearance≥ 2× institutional upper limit of normal)
* liver dysfunction not related to lymphoma(transaminase≥3× institutional upper limit of normal,and/or bilirubin≥2.0mg/dl)
* clinical syndrome of encephalon functional disorder,serious psychosis
* female subject who is pregnant or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: untreated CD20 positive Difussed large B cell lymphoma adults
Sampling Method: Probability Sample
Enrollment: 732 (Estimated)
Dates: Start 2008-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5-year

SECONDARY OUTCOMES:
5-year overall survival | 5-year
response rate | 5-year
Number of participants with SAE | 5-year
quality of life | 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Lin TongYu, Study Chair — Sun Yat-sen University
Locations (1):
- Tumor center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Huang H, Li X, Zhu J, Ye S, Zhang H, Wang W, Wu X, Peng J, Xu B, Lin Y, Cao Y, Li H, Lin S, Liu Q, Lin T. Entecavir vs lamivudine for prevention of hepatitis B virus reactivation among patients with untreated diffuse large B-cell lymphoma receiving R-CHOP chemotherapy: a randomized clinical trial. JAMA. 2014 Dec 17;312(23):2521-30. doi: 10.1001/jama.2014.15704. PMID 25514302